CLINICAL TRIAL: NCT01035489
Title: Echocardiographic Dyssynchrony in Heart Failure in CRT; Right Ventricular Apex v.s. High Posterior Septum
Brief Title: Trial in Cardiac Resynchronization Therapy (CRT): Right Ventricular Apex Versus High Posterior Septum
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Prof. Svein Faerestrand, Haukeland University Hospital, Dept. of Heart Disease, 5021 Bergen, Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/1991
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Heart Failure
Keywords: Pacemaker treatment in heart failure; Cardiac resynchronization therapy; DDD pacemakers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRT; RV apical lead placement (Active Comparator): Right ventricular apical lead placement in CRT
  Interventions: Device: CRT in heart failure; Right ventricular apex v.s. high posterior septum
- CRT; RV high posterior septum (Active Comparator): High posterior septal lead placement in CRT
  Interventions: Device: CRT in heart failure; Right ventricular apex v.s. high posterior septum

INTERVENTIONS:
Device: CRT in heart failure; Right ventricular apex v.s. high posterior septum — RV lead is randomized to either apex or high posterior septum
  Arms: CRT; RV apical lead placement
Device: CRT in heart failure; Right ventricular apex v.s. high posterior septum — RV lead is randomized to either apex or high posterior septum
  Arms: CRT; RV high posterior septum

SUMMARY:
In heart failure patients we hypothesised that right ventricular high posterior septum is superior to right ventricular apex in CRT and DDD pacemaker. In two separate trials we prospectively randomized the right ventricular lead placement to find evidence of differences in heart failure symptoms (NYHA-class), 6 minute hall walk and echocardiographic measurements of reverse remodelling and dyssynchrony.

ELIGIBILITY:
Inclusion Criteria:

* CRT:

  * LVEF < 35%
  * LVEDD > 5.5 cm
  * NYHA 3-4
  * QRS > 120 ms
  * Optimal medical treatment
  * Both CRT-pacemakers (CRT-P) and CRT combined with ICD (CRT-D)

Exclusion Criteria:

* Not fulfilling inclusion criteria or not written consensus

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic reverse remodelling and dyssynchrony | 3, 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Svein Faerestrand, MD, PhD, Principal Investigator — Faerestrand S
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Kristiansen HM, Vollan G, Hovstad T, Keilegavlen H, Faerestrand S. The impact of left ventricular lead position on left ventricular reverse remodelling and improvement in mechanical dyssynchrony in cardiac resynchronization therapy. Eur Heart J Cardiovasc Imaging. 2012 Dec;13(12):991-1000. doi: 10.1093/ehjci/jes114. Epub 2012 Jun 7. PMID 22677455
- [Derived] Kristiansen HM, Hovstad T, Vollan G, Keilegavlen H, Faerestrand S. Clinical implication of right ventricular to left ventricular interlead sensed electrical delay in cardiac resynchronization therapy. Europace. 2012 Jul;14(7):986-93. doi: 10.1093/europace/eur429. Epub 2012 Feb 2. PMID 22308084
- [Derived] Kristiansen HM, Vollan G, Hovstad T, Keilegavlen H, Faerestrand S. A randomized study of haemodynamic effects and left ventricular dyssynchrony in right ventricular apical vs. high posterior septal pacing in cardiac resynchronization therapy. Eur J Heart Fail. 2012 May;14(5):506-16. doi: 10.1093/eurjhf/hfr162. Epub 2012 Jan 26. PMID 22286156